CLINICAL TRIAL: NCT05665452
Title: Efficacy of Adding Patellar Mobilization to Hip and Knee Exercises in Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadia Abdo Mohamed Abdelhafez, Assistant lecturer at orthopedic department of faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004020
Record Dates: First submitted 2022-10-26; First posted 2022-12-27 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; strength; stretch; mobilization; release; deep friction message; retinacula
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (1) (Active Comparator): patients will receive stretch and strength exercises
  Interventions: Procedure: Patellar mobilization, retinacula release, deep friction message, stretch and strength
- Group (2) (Experimental): patients will receive stretch, strength, patellar mobilization, retinacula release and deep friction message
  Interventions: Procedure: Patellar mobilization, retinacula release, deep friction message, stretch and strength

INTERVENTIONS:
Procedure: Patellar mobilization, retinacula release, deep friction message, stretch and strength — All exercises will be performed for 30 to 45 minutes per session, 3 times per week for 4 weeks (12 sessions). Group (1): stretch exercises are performed for calf, hamstring, iliotibial band and quadriceps. strength exercises consist from open kinetic chain (hip abductors, hip external rotators and quadriceps) and closed kinetic chain exercises (mini wall squat exercise, forward step up exercise, lateral step up exercise and terminal knee extension exercise).
  Group (2): stretch exercises are performed for calf, hamstring, iliotibial band and quadriceps. strength exercises consist from open kinetic chain (hip abductors, hip external rotators and quadriceps) and closed kinetic chain exercises (mini wall squat exercise, forward step up exercise, lateral step up exercise and terminal knee extension exercise). manual therapy consists from iliotibial band release, deep friction message for lateral retinacula and medial patella mobilization.

SUMMARY:
Patellofemoral pain syndrome is a common source of anterior knee pain. The causes of PFPS may be multifactorial such as biomechanical disorders, muscle weakness which affect the dynamic stability of lower limb and alter patellar tracking in trochlear groove. Moreover, the syndrome associated with muscular tightness of iliotibial band, gastrocnemius, soleus, hamstring and quadriceps. Strengthening and stretching exercises are effective in improving patient's symptoms. However, they do not sufficient in correction of kinematic changes associated with PFPS. Patellar mobilization is effective in improving patient'symptoms in cases with PFPS. However, studies that conducted patellar mobilization were either low quality studies or no study combined patellar mobilization with hip and knee exercises.

Therefore, APTA guidelines recommended for conducting high quality study to investigate the effect of adding patellar mobilization to exercise therapy to support the definite recommendation delivered to therapists.

DETAILED DESCRIPTION:
this is interventional study in which patients will receive stretching and strengthening exercises in control group. in addition, experimental group will receive the same exercises of control group in addition to patellar mobilization, retinacula release and deep friction message.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging between 18 and 35 years
2. Tenderness of medial and lateral borders of patella
3. Retropatellar pain
4. Duration of symptoms of patellofemoral pain syndrome is greater than 4 weeks
5. Positive patellar compression test
6. Pain intensity is more than 3 at visual analogue scale
7. Had a history of insidious onset
8. Had anterior knee pain during 2 or more of provocative activities that include stair ascent or descent, kneeling, prolonged sitting, or squatting

Exclusion Criteria:

1. Previous patellar realignment surgery or patellar fracture
2. Had a history of traumatic patellar dislocation
3. Had a history of previous knee surgery
4. Had any form of inflammatory arthritis that include osteoarthritis or rheumatoid arthritis
5. Had a history of knee menisci, ligaments, bursae, or synovial plica syndrome dysfunction
6. Taking corticosteroids or nonsteroidal anti-inflammatory medication
7. Inability to attend treatment program to the end of sessions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Changes in pain that felt during ascending, descending, squatting and prolonged sitting | It will be assessed one week before and after treatment
  Pain during ascending, descending, squatting and prolonged sitting will be assessed using visual analogue scale, it is a horizontal line from 0 to 10, where 0 no pain and 10 maximum pain.
Changes in functional disability | It will be assessed one week before and after treatment
  Functional disability will be assessed using Kujala questionnaire.The scale ranges from 0 to 100 score where 100 represents no functional limitation.

SECONDARY OUTCOMES:
Changes in hip abductors strength | It will be assessed one week before and after treatment
  It will be assessed using handheld dynamometer
Changes in hip external rotators strength | It will be assessed one week before and after treatment
  It will be assessed using handheld dynamometer
changes in quadriceps strength | It will be assessed one week before and after treatment
  It will be assessed using handheld dynamometer
changes in functional performance | It will be assessed one week before and after treatment
  It will be assessed using step down test
changes in hamstring flexibility | It will be assessed one week before and after treatment
  It will be assessed using 90-90 test
changes in gastrocnemius flexibility | It will be assessed one week before and after treatment
  It will be assessed using ankle dorsiflexion range of motion
changes in knee valgus | It will be assessed one week before and after treatment
  It will be assessed using Q angle
changes in foot pronation | It will be assessed one week before and after treatment
  It will be assessed using navicular drop test

CONTACTS AND LOCATIONS:
Overall Officials: Nadia A Mohamed, Msc, Principal Investigator — Assistant lecturer at orthopedic department of faculty of physical therapy
Locations (1):
- Cairo University, Giza, Egypt

REFERENCES:
- [Derived] Abdo N, Youssef EF, Ibrahim MM. Efficacy of adding manual therapy to hip and knee exercises in patients with patellofemoral pain syndrome: a double-blinded randomized controlled clinical trial. Sci Rep. 2025 Sep 23;15(1):32655. doi: 10.1038/s41598-025-17453-9. PMID 40987761